CLINICAL TRIAL: NCT05633199
Title: Cytoreductive Surgery in Platinum-resistant Recurrent Ovarian Cancer：a Randomized Controlled Study
Brief Title: Cytoreductive Surgery in Platinum-resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPROC
Record Dates: First submitted 2022-11-20; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Cytoreductive Surgery
MeSH Terms: interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cytoreduction surgery followed by chemotherapy (Experimental)
  Interventions: Other: cytoreductive surgery
- chemotherapy alone (No Intervention)

INTERVENTIONS:
Other: cytoreductive surgery — Open surgery is conducted by senior doctors in gynecological oncology. The following parameters should be recorded: period of operation, location and number of recurrent lesions, location and number of resected lesions, amount of intraoperative bleeding and blood transfusion, whether R0 is reached, size and distribution of residual lesions, surgical complications, hospital stay, and period to adjuvant chemotherapy. Patients are required to start intravenous chemotherapy within 4W after surgery, at least for 4 cycles.
  Arms: cytoreduction surgery followed by chemotherapy

SUMMARY:
This novel study was specifically designed for platinum-resistant recurrent ovarian cancers with PFI<6 months and aimed to compare prognosis of patients who received cytoreductive surgery followed by chemotherapy versus chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of epithelial ovarian carcinoma, peritoneal carcinoma, or fallopian tube carcinoma within 3 lines recurrence;
2. Recurrence occurred within 6 months since platinum-based chemotherapy;
3. R0 ideal debulking in initial surgery; PET-CT indicate the recurrence lesion is almost in abdominal cavity, which is isolated and not exceed 5 sites, and the ascites is less than 500ml;
4. ECOG/WHO Performance score of 0 to 1;
5. Hematology function: Leukocyte≥ 3,5x10⁹/L, neutrophil≥ 1,5x10⁹/L, platelets ≥ 100x10⁹/L;
6. No Renal insufficiency: serum creatinine < 1,5 time the normal limit, creatinine clearance > 60 mL/min;
7. No hepatic failure: bilirubin ≤ 1,5 time the Normal limit;
8. Patients with good compliance;
9. Patients having read, signed and dated Informed consent before any study procedure.

Exclusion Criteria:

1. Platinum-refractory/uncontrolled epithelial ovarian cancer;
2. Mucous carcinoma or low-grade serous carcinoma;
3. Suffering from other malignant tumors that have not achieved complete remission in the past 2 years;
4. Patients have received abdominal or pelvic radiotherapy;
5. General conditions cannot tolerate cytoreduction;
6. Severe hypersensitivity reactions (≥ grade 3) to paclitaxel or platinum and/or any of its excipients;
7. Unable or unwilling to sign the informed consent form;
8. Patients judged by the investigator to be unlikely to follow the research steps, restrictions and requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | month 6
  period from the end of treatment to the recurrence of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital, Zhejiang University School of Medicine, Hangzhou, China

REFERENCES:
- [Derived] Chen T, Xu J, Xia B, Wang H, Shen Y. Evaluation of secondary cytoreduction surgery in platinum-resistant ovarian cancer patients within three-line recurrent: a multicenter, randomized controlled study. J Gynecol Oncol. 2024 Jan;35(1):e22. doi: 10.3802/jgo.2024.35.e22. Epub 2023 Oct 30. PMID 37945326